CLINICAL TRIAL: NCT04974307
Title: Pilot Study of an Optic-to-Audio Device in a Pediatric Cohort With CLN3-related Conditions or Low Vision
Brief Title: Optic-to-Audio Device in a Pediatric Cohort With CLN3-related Conditions or Low Vision
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to low enrollment
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10000414; 000414-CH
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-02

CONDITIONS: CLN3-related Disorders; Non-CLN3 Related Low Vision
Keywords: OrCam; Legal blindness; Safety; Feasibility; Efficacy
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Children with CLN3 disease (Experimental): Children with CLN3 use the OrCam MyEye 2, a 22.5-g portable, eyeglass-mounted device that converts camera-captured inputs to auditory outputs for text reading, facial recognition, and product identification. The study participants and parents/guardians were trained on how to use the device.
  Interventions: Device: OrCam MyEye 2
- Children with Low vision without CLN3 (Experimental): Children with low vision not related to CLN3 use the OrCam MyEye 2, a 22.5-g portable, eyeglass-mounted device that converts camera-captured inputs to auditory outputs for text reading, facial recognition, and product identification. The study participants and parents/guardians were trained on how to use the device.
  Interventions: Device: OrCam MyEye 2

INTERVENTIONS:
Device: OrCam MyEye 2 — The OrCam MyEye 2 is a 22.5-g portable, eyeglass-mounted device that converts camera-captured inputs to auditory outputs. Its advertised functions include text reading, facial recognition, and product identification.

SUMMARY:
Background:

CLN3 involves vision loss observed around the preschool years, with eventual progression to blindness within 1-3 years. Researchers want to test an assistive device that may help children with CLN3 or with non-CLN3 related blindness.

Objective:

To learn if it is safe, easy, and useful for children with CLN3 or with non-CLN3 related blindness to use the OrCam.

Eligibility:

People aged 6-18 years who have either CLN3-related disease or non-CLN3 related blindness.

Design:

Participants will be screened with the following:

Medical history

Physical exam

Family history

Eye exam and vision tests. They will get eyedrops to dilate their eyes.

Psychological and neurocognitive tests. They will be asked questions and observed for how they do various tasks, such as talking, playing, writing, drawing, and solving problems.

Hearing tests. They may wear headphones or earplugs. Electrodes may be taped to their head.

Blood samples

Skin biopsy, if needed

Cheek cell, saliva, or urine samples

The OrCam is the size of and weighs about half as much as a pack of gum. It is attached to eyeglass frames by magnets. Participants will do tasks before and after they have been trained on the OrCam. They will do these tasks without or with using the OrCam.

Participants will be given an OrCam to use for 1 week or 1 month. They will have check-in sessions with the study team.

Participants and/or their caregivers will be asked about abilities, behaviors, social skills, learning methods, intelligence, and health-related quality of life.

Participants samples may be used for genetic testing and/or to make a type of stem cell.

Participation will last for 1-5 weeks.

DETAILED DESCRIPTION:
Study Description:

This is a pilot study of an augmentative visual device, OrCam MyEye 2 (OrCam), in pediatric individuals with CLN3-related conditions or low vision. We hypothesize that, given the relatively simple design and operating procedure of the device, the use of the OrCam by study participants will be safe and feasible. We also hypothesize that the device will enhance their ability to obtain visually based information.

Objectives:

Primary: Assess the safety and feasibility of OrCam use by children with CLN3 or low vision.

Endpoints:

Primary:

1. Adverse events during the use of OrCam
2. Feasibility test
3. Feasibility questionnaire

The assessment periods will be 1 week at study site.

ELIGIBILITY:
INCLUSION CRITERIA:

To participate in the screening portion of this study, an individual must meet all of the following criteria:

1. Have a diagnosis or suspected diagnosis of any genetically based condition causing low vision to the level specified in criteria 2.

   If the genetic condition is CLN3-related, the individual must have one of the following:
   * a. Two CLN3 pathogenic variants, OR
   * b. One CLN3 pathogenic variant AND

     * i. clinical presentation suggestive of CLN3, OR
     * ii. characteristic electron microscopy (EM) findings (such as curvilinear body, fingerprint profile, granular osmiophilic deposits).
2. Have an estimated visual acuity in the better seeing eye < 20/200, without the use of an assistive or augmentative device.
3. Is between 6 to 18 years of age.

To participate in the intervention/device use portion of this study, an individual must meet the above screening criteria and the following criteria:

* Have an appropriate cognitive developmental ability to participate based on Investigators screening assessment.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Has any of the following auditory dysfunctions: non-reversible or non-correctable hearing loss, tinnitus that is chronic or occurring daily, auditory hallucinations that occur daily.
* Uses an optic-to-audio assistive device at the time or within 3 months of screening and enrollment.
* Is unable to travel to the NIH because of medical condition for required in-person portions of the study.
* Is unable to comply with or have medical conditions that would potentially increase the risk of participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: An N Dang Do, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie results in a publication will be shared.
Time Frame: Data may be requested 5 years after the completion of the primary endpoint
Access Criteria: Contact the principal investigator or National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000414-CH.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 11 participants consented for the study, one participant was a screen failure
Period: Overall Study
Arm/Group | Children With CLN3 Disease | Children With Low Vision Without CLN3
Started | 9 | 1
Completed | 9 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With CLN3 Disease | Children With Low Vision Without CLN3 | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 1 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: Number of participants with adverse events related to the use of OrCam MyEye 2. Adverse events were collected from parental report.
Time Frame: 1 week
Population: All participants who completed week one of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With CLN3 Disease | Children With Low Vision Without CLN3
Number analyzed (Participants) | 9 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: One week and up to one month depending on length of participation in study
Arm/Group | Children With CLN3 Disease | Children With Low Vision Without CLN3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 1/9 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children With CLN3 Disease (N=9) | Children With Low Vision Without CLN3 (N=1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination due to low subject enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04974307/Prot_SAP_000.pdf